CLINICAL TRIAL: NCT03264560
Title: Comparison of Asynchronous Telepsychiatry vs. Synchronous Telepsychiatry in Skilled Nursing Facilities: A Randomized, Controlled, Non-inferiority Trial (CATeleST)
Brief Title: Comparison of Asynchronous Telepsychiatry vs. Synchronous Telepsychiatry in Skilled Nursing Facilities
Acronym: CATeleST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1078220; 1R01HS025395 (AHRQ)
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Psychiatric Disorder
Keywords: Telepsychiatry; Synchronous; Asynchronous; SNF
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous Telepsychiatry (STP) group (Active Comparator)
  Interventions: Behavioral: Telepsychiatry
- Asynchronous Telepsychiatry (ATP) group (Experimental)
  Interventions: Behavioral: Telepsychiatry

INTERVENTIONS:
Behavioral: Telepsychiatry — A total of 6 synchronous or asynchronous telepsychiatry interventions conducted via telecommunications done at baseline, 1 month, 2 months, 3 months, 6 months, and 12 months.

SUMMARY:
There is a critical shortage of psychiatric services to people with mental illness who live in Skilled Nursing Facilities (SNFs), especially those in rural settings. Although real-time video conferencing psychiatric consultation, termed Synchronous Telepsychiatry (STP), has been around for almost 3 decades, its adaptation is met with logistic and other challenges. In this context, the investigators investigate a novel method of psychiatric consultation termed Asynchronous Telepsychiatry (ATP). The main hypotheses are that that ATP will be as clinically effective as STP, and that it will be acceptable to patients. This study aims to evaluate the comparative clinical effectiveness of ATP vs. STP in SNF population, in a 12-month non-inferiority, randomized, controlled trial.

DETAILED DESCRIPTION:
This study aims to assess the acceptability of asynchronous telepsychiatry (ATP) and synchronous (STP) in rural, Northern California Skilled Nursing Facility (SNF) population, in a 12-month randomized controlled trial.

The study will be conducted at 5 SNFs in Northern California. SNF staff will place a formal order for psychiatric consultation to the study so that the participants can receive psychiatric care via ATP or STP. Research assistants will screen each referral by reviewing inclusion and exclusion criteria based on the psychiatric referral question. To closely match real-world practice settings, STP "clinic" will be pre-scheduled for 4 hours once per month for each site. ATP participants will be interviewed by SNF staff (and videotaped with assistance from research assistant within 5 days). The video will then by reviewed by research psychiatrist and a consultation report will be send to the PCP in <5 days. Follow-up will occur at 1-, 2-, 3-, 6- and 12-month time periods, in addition to the baseline (0-month) visit for a total of 6 consults.

Aim 1: To assess whether ATP and STP models improve clinical outcomes: Hypotheses: Compared to STP, the ATP arm will: H1: show non-inferior clinical outcome trajectory, reflected in improvement from baseline, as measured by Clinical Global Impression (CGI).

Aim 2: To assess the acceptability of ATP and STP by examining satisfaction surveys from SNF residents (who are able to complete the surveys). Hypothesis: Compared to STP, ATP participants will show: H1: Similar levels of satisfaction as measured by the Telemedicine Satisfaction Survey as completed by participants.

Aim 3: To conduct healthcare economics and net benefit analysis of cost-effectiveness of ATP vs. STP in SNFs. H3: ATP, compared to STP, will be more cost effective with respect to SNF resident satisfaction and reduced wait times.

ELIGIBILITY:
Inclusion Criteria:

Participants must be residents of SNF that has been approved by University of California, Davis IRB, and adults aged ≥18, with non-emergent psychiatric issues, including:

depression, schizophrenia, bipolar disorder, PTSD, dementia behavioral problems, management of psychiatric medications, and others mental health problems. Chronic medical disorders are not excluded. Study PI or co-PI will be available by phone to help with screening.

Exclusion Criteria:

1. Residents with imminent suicidal and/or violence risks that require emergency psychiatric referrals or patients who cannot wait until the next ATP/STP evaluation,
2. Residents with imminent risks will be referred to the local emergency department as is the current practice at both SNFs, and 3) Residents who are unable to consent to the study and who do not have surrogate decisional makers to provide informed consent will not be able to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression (CGI)- severity scale | Change from baseline measure at 1-, 2-, 3-, 6- and 12-months
  Clinical outcomes from MDS 3.0 form to be collected at each consult. The primary endpoint is improvement from baseline at the 6-month visit. We will also assess long term effects of ATP, by examining 12-month outcomes.

SECONDARY OUTCOMES:
Patient Satisfaction Rating | Change from baseline measure at 1-, 2-, 3-, 6- and 12-months
  Satisfaction survey results to be collected at each consult

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/is-viewing-videotaped-interviews-with-patients-as-effective-as-psychiatric-evaluation-via-live-teleconference-in-snfs-140164/